CLINICAL TRIAL: NCT05299996
Title: Flexible URS in Management of Renal Stones in Anomalous Kidney, A Prospective Case Series Study
Brief Title: Flexible URS in Management of Renal Stones in Anomalous Kidney
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Abdelkader, principal investigator , urologist , teaching assisstant, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-URS in abnormal kidney
Record Dates: First submitted 2022-02-22; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-02

CONDITIONS: Endourology; Stones, Kidney; Laser; Congenital Disorders; Horseshoe Kidney; Malrotation of Kidney; Ectopic Kidney
MeSH Terms: conditions — Kidney Calculi; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Fused Kidney

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all patients having stones in the upper tract of anomalous kidney (Experimental): patients having stones in abnormal anatomy , example horse-shoe kidney ,malrotation, crossed fusion , duplex collecting system. The stone size is 1 cm to 2.5 cm or 3.5 cm with variable density , located in calyx or the pelvis , single or multiple.
  the patient complain may be abdominal pain , loin pain, uremic symptoms .ct-kub non contrast , full lab & fitness before the operation.
  Interventions: Procedure: flexible ureterorenoscopy

INTERVENTIONS:
Procedure: flexible ureterorenoscopy — stone disintegration stricture dilation tumor resection access guidance

SUMMARY:
The urotheliasis is a common problem encountered daily by all urologists worldwide with rates up to 13% in North America, 9% in Europe and 5% in Asia . The urotheliasis is treated by conservation, medical treatment and surgery according to many factors . Anomalies in the kidney happens due to failure in ascending , fusion, rotation or all together, horse-shoe kidney is the most common example , found in one of 400 patients . PCNL and URS are the golden standard method for stone extraction worldwide, since their introduction 1975 by Fernstrom and Johansson & Arthur Smith respectively in normal kidney .Since the development of the endourological procedures and instrument , continuous updates and upgrades have been applied ,such as enhancing the optical systems ,reducing the diameter, navigation (deflection angles) and stone fragmentation .Stone treatment in anomalous kidney is more demanding, requires more skills and training . The flexible ureterorenoscopy has some problems first the cost but this problem is being now solved by the use of disposable scopes , second the skills it requires , third the possibility of sepsis is higher . To our knowledge most of the studies in the literature are retrospective, carrying some weakness in them. There is no agreed-upon therapeutic method for treatment of stones in anomalous kidney so the investigators will evaluate the role of F-URS in a prospective study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age above 15 years.
2. Renal and ureteric stones either single or multiple wherever the site and site.
3. Pelvi-uretreic junction obstruction
4. Previous stented ureter.
5. Poorly functioning kidney.
6. Single functioning kidney.
7. Chronic kidney disease patient not on dialysis.
8. Previous operation in this kidney.
9. failed ESWL.

Exclusion Criteria:

1. Not fit for surgery.
2. Uncontrolled bleeding diathesis.
3. Untreated preoperative urinary tract infection (UTI).
4. non function kidney
5. skeletal abnormality

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
stone free rate post-operative | 1 month after treatment
  CT will be done to evaluate the presence or absence of stone
Change from Baseline hematocrit after 1 day postoperative | 1 day after treatment
  bleeding due to any error either surgical or non surgical
time of operation | during the operation
  the operation will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit Medical School, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Emiliani E, Traxer O. Single use and disposable flexible ureteroscopes. Curr Opin Urol. 2017 Mar;27(2):176-181. doi: 10.1097/MOU.0000000000000371. PMID 28027075
- [Background] Singh AG, Chhabra JS, Sabnis R, Ganpule A, Jairath A, Shah D, Desai M. Role of flexible uretero-renoscopy in management of renal calculi in anomalous kidneys: single-center experience. World J Urol. 2017 Feb;35(2):319-324. doi: 10.1007/s00345-016-1881-8. Epub 2016 Jun 15. PMID 27306685
- [Background] Giusti G, Proietti S, Peschechera R, Taverna G, Sortino G, Cindolo L, Graziotti P. Sky is no limit for ureteroscopy: extending the indications and special circumstances. World J Urol. 2015 Feb;33(2):257-73. doi: 10.1007/s00345-014-1345-y. Epub 2014 Jun 25. PMID 24962930
- [Background] Patel SR, Nakada SY. The modern history and evolution of percutaneous nephrolithotomy. J Endourol. 2015 Feb;29(2):153-7. doi: 10.1089/end.2014.0287. Epub 2014 Sep 17. PMID 25093997
- [Background] Lavan L, Herrmann T, Netsch C, Becker B, Somani BK. Outcomes of ureteroscopy for stone disease in anomalous kidneys: a systematic review. World J Urol. 2020 May;38(5):1135-1146. doi: 10.1007/s00345-019-02810-x. Epub 2019 May 17. PMID 31101967
- [Background] Alelign T, Petros B. Kidney Stone Disease: An Update on Current Concepts. Adv Urol. 2018 Feb 4;2018:3068365. doi: 10.1155/2018/3068365. eCollection 2018. PMID 29515627